CLINICAL TRIAL: NCT00000935
Title: Evaluation of Intravenous Gamma Globulin (IVIG) As an Agent to Lower Allosensitization and Improve Allograft Survival in Highly-Sensitized Adult End-Stage Renal Disease (ESRD) Patients (IG02)
Brief Title: An Evaluation of IV Gamma Globulin As a Method to Improve Kidney Transplant Survival in Patients With End-Stage Renal Disease Who Are Highly Sensitized to Transplant Antigens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT IG02
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: End-Stage Renal Disease; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Immune Globulin (Human) (Experimental)
  Interventions: Biological: Intravenous immune globulin (IVIG)
- Intravenous Immune Globulin (Human) Placebo (Placebo Comparator)
  Interventions: Biological: Intravenous immune globulin (IVIG)

INTERVENTIONS:
Biological: Intravenous immune globulin (IVIG) — given at a dose of 20mL/kg Intravenous Immune Globulin (Human) (IVIG 10% solvent/detergent)

SUMMARY:
This study is designed to test the clinical and laboratory observations that suggest IVIG given before and after kidney transplant to patients who are sensitized (highly sensitive) to certain transplant antigens could result in reduced sensitization and reduced rates of kidney rejection.

Some ESRD patients are highly sensitive to certain transplant antigens (foreign substances that activate the immune system) and must wait for a long time before a well-matched kidney becomes available. Transplant rejection is more likely among highly sensitized patients than in patients who are not highly sensitized. There is no proven method to improve a highly-sensitized patient's chances of receiving and keeping a transplanted kidney.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for patients with end-stage renal disease (ESRD). However, many patients do not receive this treatment due to immune sensitization to HLA antigens. IVIG has been shown to somewhat reduce anti-HLA antibody activity. By blocking this activity, IVIG may make transplants more feasible and increase graft survival in transplant recipients.

Patients are randomized to receive IV infusion of either 2 g/kg (maximum dose 180 g) IVIG 10% S/D (Gamimune-N, 10%, manufactured by Bayer) or placebo (0.1% human albumin, manufactured by Bayer) at time of dialysis at study entry and monthly for 3 months. If patients have not received a transplant at 1 year, they receive a "booster" dose of IVIG or placebo; patients receive another booster at 24 months if transplant still has not occurred. If transplant occurs, patients receive 2 g/kg (up to 180 g) IVIG or placebo monthly for 4 months, beginning at time of transplant. Before and after initiation of IVIG/albumin placebo treatment, specific immune parameters, including panel reactive antibodies (PRA) levels, MLR, serum inhibition of MLR, and cytokine gene transcription in the MLR, and AECA levels are measured. Outcomes studied include time on dialysis and graft survival rates.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 12 years of age or older.
* Have end-stage renal disease.
* Currently receive either hemo- or peritoneal dialysis.
* Have an elevated (> 50%) level of panel reactive antibodies (PRA level) on 3 consecutive monthly tests.
* Agree to practice sexual abstinence or to use effective means of birth control/contraception during the study and for 1 year after.

Exclusion Criteria

You will not be eligible for this study if you:

* Have received IVIG for any reason within 6 months prior to enrollment.
* Are HIV positive.
* Are Hepatitis B e-antigen/hepatitis B viral DNA-positive.
* Have selective IgA deficiency or have known antibodies to IgA.
* Are allergic to human immune globulin.
* Are pregnant or breast-feeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Penalized months of dialysis during the study | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Jordan, MD, Principal Investigator — Department of Pediatrics, Cedars-Sinai Medical Center
Locations (1):
- Ann Limberger, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY355 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY355 — ImmPort study identifier is SDY355.
- Available data/document: Study Protocol: SDY355 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY355 — ImmPort study identifier is SDY355.
- Available data/document: Study summary, -design, -demographics, -lab tests, -study files: SDY355 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY355 — ImmPort study identifier is SDY355.